CLINICAL TRIAL: NCT01972815
Title: Reproducibility and Reliability of Epstein-Barr Virus (EBV) DNA/RNA Measures in Nasopharyngeal Swabs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201205060RIB
Record Dates: First submitted 2013-10-24; First posted 2013-10-30 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Suspect NPC Patients; NPC Multiplex Families

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Nasopharyngeal carcinoma (NPC) is a virus-associated cancer that is rare among Caucasians but occurs at an elevated rate among Southern Asians. Rates of NPC are particularly high among individuals with a family history of this disease, but no specific genetic factors have been identified that can serve to guide clinical management of this high-risk population to ensure early detection and treatment of this life-threatening condition.

ELIGIBILITY:
Inclusion Criteria:

* suspect NPC patients

Exclusion Criteria:

-

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: suspect NPC patients
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-10; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
positive agreement among the positives, coefficient of variation | Four years
positive agreement among the positives, coefficient of variation | four years
  CV=SD/mean * 100

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Jen Lou, Principal Investigator — National Taiwan University Hospital
Locations (1):
- Nation Taiwan University Hospital, Taipei, Taiwan